CLINICAL TRIAL: NCT05531955
Title: A Study of Pirfenidone in the Treatment of Myocardial Fibrosis After Acute Myocardial Infarction: a Phase II Prospective, Randomized, Double-blind，Placebo Controlled Clinical Trial
Brief Title: Pirfenidone Treat Myocardial Fibrosis After Acute Myocardial Infarction
Acronym: PROTECT-AMI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHZS- F647-PIN-202201
Record Dates: First submitted 2022-08-18; First posted 2022-09-08 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Myocardial Fibrosis
MeSH Terms: interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pirfenidone group (Experimental): Drug name:Pirfenidone Dosage Form:capsule Dosage:200mg three times a day in 1st week;400mg three times a day in 2ndweek;600mg three times a day in 3rd week~52th week.
  Interventions: Drug: Pirfenidone Oral Capsule
- Placebo group (Placebo Comparator): Drug name:Placebo Dosage Form:capsule Dosage:200mg three times a day in 1st week;400mg three times a day in 2ndweek;600mg three times a day in 3rd week~52th week.
  Interventions: Other: Placebo Oral Capsule

INTERVENTIONS:
Drug: Pirfenidone Oral Capsule — pirfenidone capsules were added to patients receiving basic treatment
  Arms: Pirfenidone group
Other: Placebo Oral Capsule — placebo oral capsules were added to patients receiving basic treatment
  Arms: Placebo group

SUMMARY:
Acute myocardial infarction (AMI) is myocardial necrosis caused by acute and continuous ischemia and hypoxia of coronary artery. It can be complicated with arrhythmia, shock or heart failure, which is often life-threatening. The disease is the most common in Europe and the United States, where about 1.5 million people suffer from myocardial infarction every year. China has shown an obvious upward trend in recent years, with at least 500000 new cases every year and at least 2 million current cases . At present, China has a high incidence rate of heart failure after myocardial infarction. The incidence of heart failure within 7 days after myocardial infarction is 19.3%, and the incidence of heart failure from 30 days to 6.7 years after myocardial infarction is 13.1%~37.5%. The incidence of heart failure after myocardial infarction significantly increases the risk of short-term and long-term death, and the prognosis is poor. At present, there is a lack of unified guidance and norms for the diagnosis, treatment and prevention and control strategies of heart failure after myocardial infarction. Cardiac remodeling is the basic pathological process of heart failure after myocardial infarction, and it is also one of the main factors affecting the prognosis of patients. Studies have shown that 30% of AMI have ventricular remodeling 6 months after percutaneous coronary intervention (PCI), and the risk of ventricular remodeling in anterior wall myocardial infarction is the highest. According to foreign literature data, the probability of ventricular remodeling after anterior wall acute myocardial infarction is about 13%, which is 1.9 times higher than that in other parts.Opening the infarct related coronary artery early can save the dying myocardium, reduce the infarct myocardial area and reduce the loss of cardiomyocytes.

DETAILED DESCRIPTION:
It plays an important role in preventing or delaying the occurrence of heart failure after myocardial infarction.However,even if the blood supply of infarct related vessels is restored, the immune injury, inflammatory response and RAAS activation caused by apoptotic and necrotic cardiomyocytes after myocardial infarction will still directly lead to a series of pathophysiological changes and aggravate cardiac remodeling. Based on the above targets β Receptor blockers, ACEI / ARB / Arni and aldosterone receptor antagonists have become the cornerstone of drug therapy for cardiac remodeling after myocardial infarction. However, myocardial fibrosis also plays an important role in the process of cardiac remodeling after myocardial infarction. Ischemic death of cardiomyocytes after myocardial infarction can induce repair response, and the damaged tissue is replaced by fibrotic scar produced by fibroblasts and myofibroblasts. Although the initial reparative fibrosis is very important to prevent ventricular wall rupture, excessive fibrosis and reactive fibrosis in non infarcted areas, including myocardial interstitial and perivascular fibrosis, will cause changes in cardiac morphology and biomechanics, further aggravate cardiac remodeling, damage cardiac function, and eventually lead to heart failure. Therefore, inhibition of reactive fibrosis in non infarcted areas is an important supplement to the current treatment of traditional anti cardiac remodeling drugs. In order to reduce the degree of reactive fibrosis in non infarct areas, a potentially feasible method is to inhibit the signal pathway promoting fibrosis. TGF- β Signal pathway plays an important role in promoting fibrosis signal pathway. It can promote the proliferation of fibroblasts, the differentiation and transfer of myofibroblasts, the deposition of collagen and the survival of myofibroblasts, so it can inhibit TGF- β Signal pathway is an effective method to inhibit myocardial fibrosis.

Pirfenidone (PFD) is TGF- β The inhibitor can be used to delay the progression of idiopathic pulmonary fibrosis (IPF). Animal experiments also show that PFD can inhibit TGF- β Reduce myocardial fibrosis and improve the ability of myocardial contraction and relaxation. In the mouse model of dilated cardiomyopathy, it can effectively inhibit the pathological process of dilated cardiomyopathy, improve the degree of cardiac dilation and ventricular wall thickness. Preclinical studies have shown that PFD can inhibit myocardial fibrosis and protect the heart. A recently published phase II clinical study showed that compared with placebo, PFD significantly reduced EF value, preserved myocardial extracellular volume (ECV) and improved myocardial fibrosis in patients with heart failure (HFPEF). In view of the above background, we propose a research assumption: for patients after AMI, PFD drug intervention on the basis of standard treatment may achieve the effect of inhibiting myocardial fibrosis in non infarcted areas, so as to prevent or delay the occurrence of ventricular remodeling and heart failure after myocardial infarction, improve the quality of life and improve the prognosis of patients

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 80 years old (including 18 and 80 years old), regardless of gender.
2. Patients with acute anterior myocardial infarction 2-4 weeks after PCI.
3. NT proBNP ≥ 800 pg / ml in patients with sinus rhythm and 2400 pg / ml in patients with atrial fibrillation.
4. LVEF <50%.
5. The patients volunteered to participate in the trial, with good compliance and the ability to understand and sign the informed consent before the study

Exclusion Criteria:

1. Those who do not meet any of the inclusion criteria.
2. Patients with non acute anterior myocardial infarction.
3. Patients without PCI after myocardial infarction.
4. Glomerular filtration rate (CKD-EPI equation) < 30 ml / min / 1.73 m2.
5. Moderate or severe liver cirrhosis, or TBIL > 2 times ULN, ALT or AST > 3 times ULN caused by non cardiac reasons.
6. Patients with malignant tumors.
7. Patients with dysphagia or clinical signs of absorption disorder or requiring parenteral nutrition.
8. Patients with active peptic ulcer.
9. Severe pulmonary hypertension (pulmonary systolic pressure > 70mmhg).
10. Other diseases or complications that may affect the participation in the trial or put the patient at risk based on the judgment of the investigator.
11. Allergic to the test drug or its components (e.g., lactose).
12. Major surgery is planned during treatment.
13. Women who are pregnant, breastfeeding or planning to become pregnant during the trial.
14. Women of childbearing age are unwilling or unable to use highly effective contraceptive methods 28 days before administration or 3 months after administration.
15. According to the researchers, the patients had alcohol or drug abuse.
16. Patients with mental illness.
17. Participate in clinical trials of other drugs.
18. The researchers judged the participants who were unwell.
19. Patients who need to use Nintedanib, pirfenidone and Amifostine at the same time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Changes of the subjects'ECV | 52week
  Compare the ECV of subjects

SECONDARY OUTCOMES:
Cardiovascular death | 52week
  Number of participants with cardiovascular death
Admission for heart failure | 52week
  Number of participants for heart failure
Death | 52week
  collect the case of death
Changes of LVE | 52week
  compare the LVEF of the subjects
Changes of NT-proBNP | 52week
  compare the NT-proBNP of the subjects
Changes of ST2 | 52week
  compare the ST2 of the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Doctor, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Talman V, Ruskoaho H. Cardiac fibrosis in myocardial infarction-from repair and remodeling to regeneration. Cell Tissue Res. 2016 Sep;365(3):563-81. doi: 10.1007/s00441-016-2431-9. Epub 2016 Jun 21. PMID 27324127
- [Background] Prabhu SD, Frangogiannis NG. The Biological Basis for Cardiac Repair After Myocardial Infarction: From Inflammation to Fibrosis. Circ Res. 2016 Jun 24;119(1):91-112. doi: 10.1161/CIRCRESAHA.116.303577. PMID 27340270
- [Background] Lee HC, Park JS, Choe JC, Ahn JH, Lee HW, Oh JH, Choi JH, Cha KS, Hong TJ, Jeong MH; Korea Acute Myocardial Infarction Registry (KAMIR) and Korea Working Group on Myocardial Infarction (KorMI) Investigators. Prediction of 1-Year Mortality from Acute Myocardial Infarction Using Machine Learning. Am J Cardiol. 2020 Oct 15;133:23-31. doi: 10.1016/j.amjcard.2020.07.048. Epub 2020 Jul 26. PMID 32811651
- [Background] Dondo TB, Hall M, Munyombwe T, Wilkinson C, Yadegarfar ME, Timmis A, Batin PD, Jernberg T, Fox KA, Gale CP. A nationwide causal mediation analysis of survival following ST-elevation myocardial infarction. Heart. 2020 May;106(10):765-771. doi: 10.1136/heartjnl-2019-315760. Epub 2019 Nov 15. PMID 31732655
- [Background] Lewis GA, Dodd S, Clayton D, Bedson E, Eccleson H, Schelbert EB, Naish JH, Jimenez BD, Williams SG, Cunnington C, Ahmed FZ, Cooper A, Rajavarma Viswesvaraiah, Russell S, McDonagh T, Williamson PR, Miller CA. Pirfenidone in heart failure with preserved ejection fraction: a randomized phase 2 trial. Nat Med. 2021 Aug;27(8):1477-1482. doi: 10.1038/s41591-021-01452-0. Epub 2021 Aug 12. PMID 34385704
- [Background] Graziani F, Lillo R, Crea F. Rationale for the Use of Pirfenidone in Heart Failure With Preserved Ejection Fraction. Front Cardiovasc Med. 2021 Apr 22;8:678530. doi: 10.3389/fcvm.2021.678530. eCollection 2021. PMID 33969025
- [Background] Lewis GA, Schelbert EB, Naish JH, Bedson E, Dodd S, Eccleson H, Clayton D, Jimenez BD, McDonagh T, Williams SG, Cooper A, Cunnington C, Ahmed FZ, Viswesvaraiah R, Russell S, Neubauer S, Williamson PR, Miller CA. Pirfenidone in Heart Failure with Preserved Ejection Fraction-Rationale and Design of the PIROUETTE Trial. Cardiovasc Drugs Ther. 2019 Aug;33(4):461-470. doi: 10.1007/s10557-019-06876-y. PMID 31069575
- [Background] Nguyen DT, Ding C, Wilson E, Marcus GM, Olgin JE. Pirfenidone mitigates left ventricular fibrosis and dysfunction after myocardial infarction and reduces arrhythmias. Heart Rhythm. 2010 Oct;7(10):1438-45. doi: 10.1016/j.hrthm.2010.04.030. Epub 2010 Apr 28. PMID 20433946
- [Background] Li C, Han R, Kang L, Wang J, Gao Y, Li Y, He J, Tian J. Pirfenidone controls the feedback loop of the AT1R/p38 MAPK/renin-angiotensin system axis by regulating liver X receptor-alpha in myocardial infarction-induced cardiac fibrosis. Sci Rep. 2017 Jan 16;7:40523. doi: 10.1038/srep40523. PMID 28091615